CLINICAL TRIAL: NCT04283305
Title: A Randomized Controlled Trial of a Virtual Reality Based, Approach-avoidance Training Program for Alcohol Use Disorder
Brief Title: Virtual Reality Alcohol Avoidance Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Odense University Hospital (Other); Pomeranian Medical University Szczecin (Other); European Regional Development Fund (Other); Hochschule für Techink und Wirtschaft Berlin (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VR_AAT
Record Dates: First submitted 2020-02-14; First posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Alcohol Use Disorder
Keywords: approach bias; virtual reality; training
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of three conditions:
  1. = virtual reality approach avoidance training
  2. = computer-based approach avoidance training
  3. = treatment as usual
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual reality approach avoidance training (Experimental): Participants will receive six sessions (three sessions per week for two weeks; session duration = 30 mins) of approach-avoidance training in the virtual reality. Alcoholic beverages are pushed away with a controller and soft-drinks will be pulled towards oneself. Training will begin approximately three weeks before discharge from the inpatient clinics to measure the add-on effect and to ensure that the add-on treatment does not extend the treatment period.
  Interventions: Other: Virtual reality approach avoidance training
- Computer-based approach avoidance training (Active Comparator): Participants will receive six sessions (three sessions per week for two weeks; session duration = 30 mins) of approach-avoidance training on the computer. Alcoholic beverages are pushed away with a joystick and soft-drinks will be pulled towards oneself. Training will begin approximately three weeks before discharge from the inpatient clinics to measure the add-on effect and to ensure that the add-on treatment does not extend the treatment period.
  Interventions: Other: Computer-based approach avoidance training
- Treatment as usual (No Intervention): Participants will receive treatment as usual on the wards. For ethical reasons, participants in this condition will get the offer to undertake the already scientifically validated computer-based approach avoidance training after their completion of the study.

INTERVENTIONS:
Other: Virtual reality approach avoidance training — In the VR-based AAT, patients are situated in a bar environment where drinks appear on a bar table in front of them. Patients are instructed to react to 100% of the alcoholic beverages with a push response with a controller, and to non-alcoholic drinks in 100% of the trials with a pull response. The stimuli set consists of 50 different beverages, which are displayed three times in total.
  Arms: Virtual reality approach avoidance training
Other: Computer-based approach avoidance training — In the computer-based AAT, patients are situated in front of a computer where drinks appear on the screen in front of them. Patients are instructed to react to 100% of the alcoholic beverages with a push response with a joystick, and to non-alcoholic drinks in 100% of the trials with a pull response. The stimuli set consists of 50 different beverages, which are displayed three times in total.
  Arms: Computer-based approach avoidance training

SUMMARY:
The approach-avoidance training program (AATP) has shown preliminary promise as an add-on to standard treatment for alcohol dependence. However, knowledge is lacking as to whether the effectiveness of AATP can be enhanced further when performed in a typical drinking situation. The main aim of this study is to investigate whether approach-avoidance training implemented in a virtual reality bar environment is superior to the classical joystick PC-version of the AATP.

DETAILED DESCRIPTION:
The study will be implemented as a randomized controlled trial. A total of 135 consecutively enrolled alcohol use disorder (AUD) patients, recruited from alcohol inpatient clinics in Germany, Poland and Denmark, will be randomized into one of three groups at the start of standard alcohol treatment: group A) stimuli-relevant AATP as usual; group B) stimuli-relevant ATTP in virtual reality, and group C) treatment as usual (TAU; control group). Treatment outcomes will be assessed at pre-treatment, post-treatment and 3-month follow-up. Generalized mixed-models will be applied to compare the trajectories of the groups over time on drinking, craving and impulsiveness outcomes.

ELIGIBILITY:
Inclusion Criteria:

* signed written informed consent
* meeting the diagnostic criteria for alcohol use disorder
* fluent in language of the participating country (German, Polish or Danish)
* completion of detoxification (if needed)
* enrolled in standard treatment within two weeks

Exclusion Criteria:

* any sensory or motor deficits complicating the provision of the AAT (e.g. color-blindness, fine or gross motor deficits in upper extremities)
* meeting diagnostic criteria for other substance use disorders
* severe psychiatric or neurological illness (e.g. psychotic disorders, mental retardation, dementia) or terminal somatic illness

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 135 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Changes in alcohol consumption | at baseline (day 0), at post-test (right after 14 days training period) and at follow up (84 days after post-test)
  Alcohol consumption measures will be derived from the Timeline Followback (TLFB). The TLFB method involves using a calendar to identify alcohol consumption patterns in terms of number of drinks per day during the last 30 days. One drink is defined as 12 grams of ethanol. The Visual Analogue Scale (VAS) comprises single items used to measure the degree of alcohol cravings on scales ranging from 0-100, with 0 representing no cravings and 100 an extreme degree of cravings. The scale is presented visually on a ruler, and the individual will be requested to report the frequency, mean level and the peak level of cravings experienced during the last 30 days.

SECONDARY OUTCOMES:
Changes in alcohol-related craving | at baseline (day 0), at post-test (right after 14 days training period) and at follow up (84 days after post-test)
  The 14-item obsessive-compulsive drinking scale (OCDS) measures the degree of cravings experienced during the last seven days. Items are rated on scales ranging from 0 to 4. The higher the score, the more pronounced the cravings. The scale has two subscales: obsessive cravings score and compulsive cravings score. A total score is calculated based on these subscales, and it is possible to calculate a resistance/impairment and interference subscale score.
Changes in alcohol abstinence self-efficacy | at baseline (day 0), at post-test (right after 14 days training period) and at follow up (84 days after post-test)
  The 40-item Alcohol Abstinence Self-Efficacy Scale (AASE) measures current level of temptation to drink alcohol and self-efficacy to abstain from drinking. The scale applies 20 situations representing typical drinking cues. Twenty items pertain to temptation levels, the other 20 items to self-efficacy. Items are rated on scales ranging from not at all (0) to extremely (4). The measure comprises the following sub-scales: (1) negative affect; (2) social interaction and positive states; (3) physical and other concerns; and (4) withdrawal and urges (40).
Changes in impulsivity | at baseline (day 0), at post-test (right after 14 days training period) and at follow up (84 days after post-test)
  The 30-item Barratt impulsiveness scale (BIS, Patton, Stanford, & Barratt, 1995) assesses dimensions of impulsivity using three subscales: (1) attentional (attention and cognitive instability), (2) motor (motor and perseverance); and (3) non-planning (self-control and cognitive complexity). Items are rated on 4-point Likert scales ranging from 1 = very true for me to 4 = very false for me.
Changes in depression severity | at baseline (day 0), at post-test (right after 14 days training period) and at follow up (84 days after post-test)
  The Beck Depression Inventory-II (BDI-II; Beck et a., 1996) is a 21-item multiple-choice instrument that measures the severity of depression. Each item is rated on a 4-point scale ranging from 0 to 3 based on severity.

OTHER OUTCOMES:
Changes in Alcohol related Approach Bias | at baseline (day 0), at post-test (right after 14 days training period) and at follow up (84 days after post-test)
  The diagnostic alcohol-approach-avoidance task (alcohol-AAT) measures approach biases. During the alcohol- AAT, AUD individuals are requested to react to pictures of alcoholic and non-alcoholic drinks using approach and avoidance responses (by pulling or pushing a joystick (comuter-based AAT) or a controller (VR-AAT)). 50% of the alcoholic/non-alcoholic beverages are pushed away and 50% pulled towards oneself. An approach bias is indicated when reaction times are faster for approaching alcohol cues than for avoiding them, whereas the opposite indicates avoidance bias.
Changes in cue-induced cravings | at baseline (day 0), at post-test (right after 14 days training period) and at follow up (84 days after post-test)
  Cravings will be assessed for all alcoholic and non-alcoholic beverages from the conventional and VR-based AAT. The pictures will be rated on the VAS scale ranging from 0-100 according to the immediate level of craving induced to examine their potential to elicit cue-induced cravings.
Changes in alcohol-related response inhibition | at baseline (day 0), at post-test (right after 14 days training period) and at follow up (84 days after post-test)
  Response inhibition towards alcohol cues will be recorded using a modified version of the classical Go/No-Go Task. The modification involves the use of alcohol-related and neutral pictures to specifically test inhibition capacities towards alcohol-related cues. Pictures of alcoholic and non-alcoholic drinks from the conventional and VR-based AAT as well as new pictures will be included in the task. Patients will be instructed to respond as fast as possible, and without errors, by pressing a response button when they see a non-alcoholic drink (i.e. "Go" signals) but to withhold their response when an alcoholic drink is presented (i.e. "NoGo" signals).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mellentin AI, Nielsen AS, Ascone L, Wirtz J, Samochowiec J, Kucharska-Mazur J, Schadow F, Lebiecka Z, Skoneczny T, Mistarz N, Bremer T, Kuhn S. A randomized controlled trial of a virtual reality based, approach-avoidance training program for alcohol use disorder: a study protocol. BMC Psychiatry. 2020 Jun 30;20(1):340. doi: 10.1186/s12888-020-02739-1. PMID 32605614